CLINICAL TRIAL: NCT05273346
Title: Traditional Chinese Medical Comprehensive Conservative Treatment for the Degenerative Lumbar Spinal Stenosis
Brief Title: TCM Conservative Treatment for the Degenerative Lumbar Spinal Stenosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Changhe Yu, Clinical professor, Beijing University of Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021DZMEC-123-02
Record Dates: First submitted 2022-02-07; First posted 2022-03-10 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Degenerative Lumbar Spinal Stenosis
Keywords: low back pain; leg pain; Spinal Stenosis
MeSH Terms: conditions — Low Back Pain; Spinal Stenosis | interventions — Acupuncture Therapy; Cupping Therapy; Electric Stimulation Therapy; Acetaminophen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This trial is an open study. Subjects and physicians are not blinded, but outcome evaluators and statisticians are blinded. Doctors not involved in patient grouping and treatment will be appointed to evaluate the efficacy of patients. After locking the database, the third party statisticians who do not know the grouping should analyze it.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comprehensive Conservative TCM Treatment Group (Experimental): 1. Traditional Chinese medicinal ointment;
  2. Acupotomy;
  3. Cupping therapy with bamboo cup;
  4. Oral Chinese medicine granules.
  Interventions: Behavioral: Traditional Chinese medicinal ointment; Behavioral: Acupotomy; Behavioral: Cupping therapy with bamboo cup; Other: Oral Chinese medicine granules
- Modern Medicine Conservative Treatment Program Group (Active Comparator): 1. Epidural Steroid Injections (ESIs);
  2. Interferential current therapy;
  3. Thermal therapy;
  4. Oral painkillers.
  Interventions: Behavioral: Epidural Steroid Injections (ESIs); Behavioral: Interferential current therapy; Behavioral: Thermal therapy; Other: Oral painkillers

INTERVENTIONS:
Behavioral: Traditional Chinese medicinal ointment — The Group1 will be treated using the Comprehensive Conservative TCM Treatment Group protocol.The special TCM ointment will be applied to the waist, and then Tuina, in order to play the comprehensive therapeutic role of Tuina and medicine, promoting blood circulation and removing stasis, warming and dispersing cold, strengthening tendons and strengthening bones, regulating qi and blood. The method of ointment is generally used with rubbing method, rubbing method, flat pushing method and kneading method. Treatment time: 7 minutes.
  Arms: Comprehensive Conservative TCM Treatment Group
Behavioral: Acupotomy — It is in the special acupoints or Ashixue for cutting, stripping and other different stimulation, in order to reduce the tension of soft tissue outside the spinal canal, reduce the trend of dynamic and static spinal canal stenosis, to achieve the purpose of relieving pain and removing disease, opening points and collaterals. Acupotomy can separate the adhesive tissue, which can improve the blood circulation of the local tissue and promote the absorption of inflammation. Most acupotomy points are tenderness points or induration points, such as yaojiaji and Shenshu. Treatment time: 3 minutes.
  Arms: Comprehensive Conservative TCM Treatment Group
Behavioral: Cupping therapy with bamboo cup — Put the bamboo cup with the thickness of the thumb into the cup and boil it, then find the meridian and select the acupoint, Pierce the skin with a needle at the appropriate acupoint, and remove the heated bamboo cup from the cup while it is hot. When the temperature of the steam in the bamboo cup is reduced, steam will condense into water quickly, which produces strong negative pressure. Through the medicinal force, heat and the suction of the bamboo cup, the blood stasis in the affected area is smoothly discharged, so that qi and blood can be unblocked and pain can be eliminated. Treatment time: 20 minutes.
  Arms: Comprehensive Conservative TCM Treatment Group
Other: Oral Chinese medicine granules — Oral Chinese medicine granules use to nourish liver and kidney, improve qi and blood. Patients voluntarily take it when they think it is necessary.
  Arms: Comprehensive Conservative TCM Treatment Group
Behavioral: Epidural Steroid Injections (ESIs) — The Group2 will be treated using the Modern Medicine Conservative Treatment Program Group protocol.All Epidural Steroid Injections(ESIs) will be performed by a physician in an outpatient surgical setting(a sterile operating room),the patient will be in prone position,while monitored the vital signs. After aseptic treatment, 1mg non-granular betamethasone plus 5mL 0.9% sodium chloride solution will be injected. Patients will repeat ESIs up to four times within three months after randomization, depending on the response to the previous ESIs, when the degree of pain increases or the degree of relief is less than 50%.
  Other Names: ESIs
  Arms: Modern Medicine Conservative Treatment Program Group
Behavioral: Interferential current therapy — The 30-50cm padded electrode will be properly fixed on the left and right sides of the lumbar spinal stenosis, and the two groups of current will be crossed at the lesion. Constant frequency output 90Hz, frequency conversion output 90-100Hz, the current intensity is generally suitable for patient tolerance, each treatment for 10min, a total of 20 minutes. Twice a week for 3 months.
  Arms: Modern Medicine Conservative Treatment Program Group
Behavioral: Thermal therapy — After the interferential current therapy, the patient will receive Bohm light for 5 minutes at the site of lumbar spinal stenosis and massage for 5 minutes at low back. Twice a week for 3 months.
  Arms: Modern Medicine Conservative Treatment Program Group
Other: Oral painkillers — NSAID drugs, if necessary.
  Arms: Modern Medicine Conservative Treatment Program Group

SUMMARY:
Lumbar degenerative disease is a common disease develops into degenerative lumbar spinal stenosis(DLSS)in the elderly and eventually. The long course of disease and other characteristics determine that conservative treatment cannot be effective in a short time, surgery is recommended to relieve symptoms quickly. However, the incidence of complications and disease recurrence rate after surgical treatment is high, and the reoperation rate is as high as 30-50%. Conservative treatment has the advantages of low price and high acceptance, so the treatment strategy first returns to conservative treatment.The complexity and repeatability of DLSS are the main reasons for the adoption of comprehensive treatment in modern medicine, but the efficacy is not significant. Traditional Chinese medicine (TCM) has its own theories and various methods to treat low back pain.

DETAILED DESCRIPTION:
Under the guidance of TCM holistic view and syndrome differentiation views, the treatment group invented the concept of treating with tendon instead of bone and miscellaneous combination, and initially formed a four-dimensional integrated TCM comprehensive conservative diagnosis and treatment plan of moderate and severe DLSS, which is mainly composed of cupping therapy with bamboo cup, assisting with acupotomy, repairing with Traditional Chinese medicinal ointment and regulating body with Chinese herb decoction. Based on evidence-based evidence, this study optimized and verified the comprehensive plan of TCM, and finally formed the technical specification, so as to enrich and improve DLSS conservative diagnosis and treatment technology, provide clinical evidence of comprehensive plan of TCM, and improve the ability of TCM to treat difficult and serious diseases. Based on the above,the investigators will carry out a randomized controlled trial (RCT) to verify the effectiveness and safey of TCM comprehensive conservative treatment. A total of 94 patients with moderate to severe DLSS were included and randomly assigned to the experimental group and the control group according to 4:3, including 53 patients in the experimental group and 41 patients in the control group. The experimental group received the comprehensive conservative treatment for 3 months, the control group accepted the modern comprehensive medical conservative treatment, treatment for 3 months, main efficacy outcome indicators for 3 months, 15 months after random based on efficient Zurich Claudication questionnaire(ZCQ), secondary outcome indicators including pain rating scale, SF-12 questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic of Degenerative Lumbar Spinal Stenosis.
* Males and females aged between 40 and 85.
* Low back pain and leg pain accompanied by typical neurogenic intermittent claudication symptoms, lasting ≧3 months.
* The effect of 3 months conservative treatment(Oral painkillers + any 1 physical therapy) was not ideal(Less than 50% relief from pain or functional limitations).
* Having any of the following surgical indications: 1.Low back and leg pain after exercise, affecting life and work (the patient felt seriously affecting life and work);2. Progressive claudication(Continuous walking distance is less than 100m),or standing time is decreasing(Standing time at a time reduced to 50% of the onset);3. Those with obvious neurological defects(Suddenly appear the paresthesia of the distribution area of spinal nerve, such as numbness, acid bilges, acupuncture feeling, limb hair cool).
* The patient refused surgical treatment.
* Willing to participate in this study, and signed the informed consent.

Exclusion Criteria:

* Patients with vasogenic intermittent claudication.
* Patients with other bone and joint diseases, including spinal vertebra fracture, lumbar tuberculosis, spinal tumor and other lesions, or rheumatism, rheumatoid arthritis.
* Patients with hematopoietic system(anemia,aplastic anemia), cardiocerebral vascular system(History of cerebral hemorrhage, Serious cardiovascular disease), endocrine system(Poor glycemic control in diabetes, such as postprandial blood glucose over 12mmol/L) and other serious primary diseases, tumors and psychosis.
* Patients with scoliosis >15° or disc instability (rotation >10° or translation >4mm).
* Patients after minimally invasive surgery and open surgery.
* Patients who received an epidural steroid injection within 6 months.
* The patient is allergic to Traditional Chinese medicine, history of skin allergy and allergic constitution.
* The treatment site has subcutaneous unknown lump, the skin is red and swollen broken ulceration inflammation or skin lesions, etc.
* Patients with severe cauda equina syndrome.
* Women who are menstruating, pregnant or breastfeeding.
* Patients with strong preferences for treatment, disobedience to random assignment, and poor compliance.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The short-term response rate | The 3rd month
  The NASS guidelines recommend the use of response rate as the primary criterion for determining performance due to the variety, complexity and repeatability of DLSS performance. The Zurich Claudication Questionnaire (ZCQ) is considered by the North American Spine Association (NASS) to be the best and most specific assessment method. It is the "gold standard" to evaluate the function of patients with lumbar spinal stenosis. Therefore, as the standard for calculating effective rate in this study, the decrease of symptom severity subscale and physiological function subscale score ≥0.5 points represents "success". A decrease of ≥2.5 points in the satisfaction subscale represents "success". When at least two subscales are judged to be "successful", the treatment is judged to be effective, thus the response rate is calculated.In ZCQ, the greater the difference between the two measurements before and after (the lower the score of the latter measurement), the better degree of recovery.
The long-term response rate | The 15rd month
  Using the Zurich Claudication Questionnaire (ZCQ) as the standard for calculating response rate in this study, the decrease of symptom severity subscale and physiological function subscale score ≥0.5 points represents "success". A decrease of ≥2.5 points in the satisfaction subscale represents "success". When at least two subscales are judged to be "successful", the treatment is judged to be effective, thus the response rate is calculated.In ZCQ, the greater the difference between the two measurements before and after (the lower the score of the latter measurement), the better degree of recovery.

SECONDARY OUTCOMES:
Changes in pain level | The time points of evaluation were baseline, 3,6,9,12 and 15 months.
  The severity of leg pain and low back pain within 24 hours was assessed by the Digital Pain Scale (NRS).10 is the highest score, indicating unbearable pain. 0 is the lowest score, meaning no pain.The higher the NRS score, the more intense of the pain.
Changes in general health status | The time points of evaluation were baseline, 3,6,9,12 and 15 months.
  Chinese version of SF12 was used to evaluate the overall health status, including total physical health score and total mental health score.After the formula score calculation, the higher the score, the better the health.
Changes in locomotor function | The time points of evaluation were baseline, 3,6,9,12 and 15 months.
  The Oswestry Disability Index (ODI) consists of 10 items, including pain, individual disability and general disability. The lowest score for each item is 0, and the highest score is 5, with higher scores indicating higher levels of dysfunction. After the corresponding scores of the answers of the 10 items are accumulated, the percentage of the answers to the highest total score (50 points) is calculated, which is ODI. The higher the score is, the more serious the patient's dysfunction is.
Incidence of surgery | The evaluation time point was 3,6,9,12, and 15 months.
  The incidence of patients attending surgical treatment was recorded at any time.

CONTACTS AND LOCATIONS:
Overall Officials: Changhe Yu, Principal Investigator — Beijing University of Chinese Medicine affiliated Dongzhimen Hospital
Locations (1):
- Dongzhimen hospital affiliated to Bejing University of Chinese Medicine, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No